CLINICAL TRIAL: NCT04575246
Title: Predictors and Outcomes of Intraoperative Hypothermia in Patients Undergoing Total Knee Arthroplasty: A Retrospective Cross-sectional Study From a Developing Country
Brief Title: Predictors and Outcomes of Intraoperative Hypothermia in Patients Undergoing Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Anum Sadruddin, Research Associate, Aga Khan University
Other Study IDs: 2019-1274-3270
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Knee Arthroplasty, Total; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is designed to retrospectively assess the risk factors associated with intra-operative hypothermia in patients undergoing total knee arthroplasty from January 2016 to December 2017 at Aga Khan University and also understand it's impact on post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All adults greater than 18 years who underwent total knee arthroplasty.

Exclusion Criteria:

* Any patient below 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults greater than 18 years undergoing total knee arthroplasty from January 2016 to December 2017 at Aga Khan University were included in this study. A standardized proforma was used to collect data from online patient data system about patients' preoperative, intraoperative and postoperative details. Preoperative data included age, gender, and comorbid conditions. Intraoperative data was collected from the surgical and anaesthesia records and included surgical site, American Society of Anesthesiologists (ASA) Level, duration of surgery, preoperative body temperature, intraoperative body temperature and duration of surgery. Postoperative data included post-operative body temperature and whether the patient developed any surgical site infection.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | 2016-2017
  Post-operative infection caused total knee arthroplasty
Post-operative hypothermia | Within an hour after surgery
  Body temperature after surgery when patient is in the recovery room.

REFERENCES:
- [Derived] Ukrani RD, Arif A, Sadruddin A, Hasan O, Noordin S. Intraoperative hypothermia in patients undergoing Total knee arthroplasty: a cross-sectional study from a developing country. BMC Musculoskelet Disord. 2021 May 31;22(1):504. doi: 10.1186/s12891-021-04390-7. PMID 34059046